CLINICAL TRIAL: NCT06957041
Title: Effect of Intertransverse Process Block on the Quality of Recovery Post-Open Hepatectomy: A Pilot Non-Randomised Study of Intervention
Brief Title: Intertransverse Process Block for Quality of Recovery Post-Open Hepatectomy
Acronym: ITPB QoR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Wing Sum Li, Resident, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRE Ref. No. 2024.562
Record Dates: First submitted 2025-04-18; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Hepatectomy; Intertransverse Process Block; Quality of Recovery (QoR-15)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open Hepatectomy Patient receiving the intertransverse process block (Experimental)
  Interventions: Procedure: Intertransverse process block

INTERVENTIONS:
Procedure: Intertransverse process block — The patient(s) will receive a pre-induction Intertransverse process block as pilot study

SUMMARY:
The study aims to assess the analgesic efficacy of the ITPB at the retro-SCTL space in patients undergoing major open hepatectomy surgery. This is assessed by:

Primary Objective:

Primary outcome measure:

● Assessing the quality of recovery 15 (QoR15) score at 24 and 48 hours

Secondary outcome measure:

* Number of anaesthetic and hypoesthetic dermatomes on the ventral and dorsal aspect of the thorax on both the sides at 30 minutes of block completion and during the post anaesthetic room (PACU) discharge
* Assessing the 24-hour area under the curve of postoperative pain numerical rating score (NRS, 0-10) at rest and deep breathing or upon use of triflow.
* Assessing the amount of postoperative morphine (mg) equivalent consumption at 24 and 48 hours
* Time to discharge from High dependency unit (HDU) or Intensive care unit (ICU)

Hypothesis:

The investigators hypothesize that the application of ITPB targeting the retro-SCTL space in patients undergoing open hepatectomy will improve overall quality of recovery and pain score.

ELIGIBILITY:
Inclusion Criteria:

- Adult patients aged 18-75 years of ASA I - III physical status classification undergoing open hepatectomy for benign or malignant liver lesion.

Exclusion Criteria:

* Patient refusal
* Patients who are unable to comprehend the QoR15 form
* Local or systemic infection
* Coagulopathy leading to absolute contraindication to regional anesthesia
* Contraindication to local anaesthetics (LA) such as LA allergy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Quality of Recovery (QOR-15) | 24 and 48 hours
  The QoR-15 scale is a global measure of postoperative recovery, with a score ranging from 0 (extremely poor QoR) to 150 (excellent QoR). The QoR-15 has since become the most widely reported measure of patient-assessed QoR after surgery. QoR-15 has no units.

SECONDARY OUTCOMES:
Dermatomal blockade on Thorax 30 minutes upon block completion | Up to 30 minutes after block completion
  To assess the number of anaesthetic and hypoesthetic dermatomes on the ventral and dorsal aspect of the thorax on both the sides at 30 minutes of block completion and during the post anaesthetic room (PACU) discharge. This will be done by ice block test. The blockade is considered positive if patient has a reduction in cold sensation over the tested dermatome compared to non-blocked areas such as forehead.
24 hours area under curve of postoperative pain score | Up to 24 hours
  Assessing the 24-hour area under the curve of postoperative pain numerical rating score (NRS, 0-10) at rest and deep breathing or upon use of triflow.
Morphine consumption at 24 and 48 hours postoperatively | At 24 and 48 hours postoperatively
  Assessing the amount of postoperative morphine (mg) equivalent consumption at 24 and 48 hours
Time to discharge from HDU / ICU | Up to 5 days
  Time to discharge from High dependency unit (HDU) or Intensive care unit (ICU) up to 5 days

IPD SHARING:
Plan to Share IPD: Undecided